CLINICAL TRIAL: NCT02643745
Title: Nephrologic Intervention in Patients Waiting for Cardiac Surgery
Acronym: AKIIcor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Nuria Montero, Dr., Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AKIIQcor
Record Dates: First submitted 2015-03-25; First posted 2015-12-31 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: ACUTE KIDNEY INJURY
Keywords: acute kidney injury; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nephrology Intervention (Experimental): Nephrology intervention before surgery:
  Interventions: Procedure: Nephrology Intervention
- Standard of Care (No Intervention): No nephrology intervention before surgery (standard of care)

INTERVENTIONS:
Procedure: Nephrology Intervention — 1. pre-operative study:
     * Kidney function: creatinine, Glomerular filtration rate (GFR) and presence albuminuria or proteinuria. Assessment whether there is a functional component added.
     * Discard presence of renal disease: renovascular disease, glomerular disease, toxic, etc.
  2. optimise the patient' s overall condition with a pre-operative strategy:
     * Obesity control
     * Control protein, caloric, salt intake
     * Stop smoking
     * Good glycemic control
     * Start ACEI/ARA II if there is proteinuria
     * Start additional antihypertensive drug if required
     * Start hypolipemic treatment if required
     * Start hyperuricemia treatment if required
     * Start AAS, clopidogrel if it is necessary (prophylaxis)
     * Phosphate control
     * Anemia control
     * Metabolic acidosis correction
  Arms: Nephrology Intervention

SUMMARY:
Acute kidney injury (AKI) is a frequent complication after cardiac surgery. Its incidence ranges from 19 to 44% depending on the study and which definition is used: Acute Kidney Injury Network (AKIN) classification or RIFLE criteria (Risk, Injury, Failure, Loss, End-Stage Kidney Disease) based on serum creatinine and urine output.

AKI is associated with increased mortality, more complications, a longer stay in the intensive care unit and hospital, and increased health care costs. Moreover, the patients who require renal replacement therapy (RRT) have the highest mortality and complications1.The mortality risk in patients developing acute renal dysfunction after cardiac surgery increases by approximately 40%, while the overall mortality rate after cardiac surgery ranges between 2% and 8%.

There are some well-known risk factors associated with AKI, including baseline patient characteristics (age and comorbidities), need of perioperative blood transfusion or presence of previous chronic kidney disease. The main objective of this study is to evaluate if a nephrologist management and control of potential risk factors of renal disease can be used to prevent AKI, thereby minimizing the risk of need RRT, reducing costs and improving survival in this patients.

DETAILED DESCRIPTION:
Aim The aim of this study is to assess if a nephrology intervention before cardiac surgery can reduce the postoperative incidence of AKI (Acute Kidney Injury).

Methods Trial design and participants Recruitment: unicentric Ethics approval: Clinical Research Ethics Committee of Bellvitge will have approved the study before initiation. All patients will give written informed consent. Patients will be able to withdraw informed consent.

Duration of the study: 3 years recruitment, 1 year follow-up.

Randomization

Eligible patients will be randomly assigned by using sequentially numbered, opaque, sealed envelopes. Patients will be allocated to one of two groups using shuffled envelopes at the moment of the first visit of the cardiac surgeon. The two groups will be:

1. Nephrology intervention before surgery, which will include:

   1. pre-operative study:

      * Kidney function: creatinine, Glomerular Filtration Rate (GFR) and presence albuminuria or proteinuria. Assessment whether there is a functional component added.
      * Discard presence of renal disease: renovascular disease, glomerular disease, toxic ...
   2. optimise the patient' s overall condition with a pre-operative strategy:
2. No nephrology intervention before surgery (standard of care) Treatment allocation will be know by the clinician entering the patient into the trial at the moment the envelope will be opened.

Blinding Open study. If it appears a clinical situation that force the clinician to change the patient allocation group (e.g. acute kidney injury or advanced chronic kidney disease not known before which requires some treatment), an intention-to-treat analysis will be made considering the results of the patient in the initial assigned group.

Procedures

Baseline data recorded:

* Age
* Race/ethnicity
* Gender
* Body mass index
* Comorbidities: coronary heart disease, previous cardiac arrest, diagnosed hypertension, cerebrovascular disease, peripheral vascular disease, diabetes type I or II, chronic obstructive pulmonary disease, cancer, inability to ambulate or transfer.
* Day of randomisation and the day on admission to hospital: serum creatinine, proteinuria (albuminuria, urine albumin-to-creatinine ratio (ACR), and protein-to-creatinine ratio (ACR), urinary ionogram, ferritin, transferrin saturation index, albumin, prealbumin, cholesterol levels (LDL, HDL, total), uric acid, fibrinogen, fasting blood glucose, HbA1c, phosphate, hemoglobin and venous blood gasometry
* Type of surgery
* Date of intervention and surgeon
* Treatment before surgery (ACEI, ARA II, non steroid antinflamatories, betablockers, statins..)
* Ejection fraction, PAP, diastolic disfunction and left ventricular dysfunction
* Postoperative need of pacemaker
* Euroscore index and index of Charlson

Operative factors:

* off-pump surgery
* clamp time (minutes)
* hemodynamic constants (medium arterial pressures)
* fluid balance
* need of blood transfusions
* number of cardioversion Patients will be followed up until they meet the primary endpoint, or for a minimum of one year if they do not do so. The trial will not formally be analyzed until 1 year after all patients will have been randomized. Follow-up information will be obtained from consultant intensivist and consultant nephrologist.

Follow up: Clinical and analytical assessment will be carried out at discharge, 4 and 12 months after surgery by the cardiac surgeon and nephrologist.

Sample size: The number of participants required in each group is calculated with 80% power and 5% significance: 9

•n= 550 per group --> considering a difference of 5% in people presenting AKI between people without nephrologist intervention before surgery (12,2%) and those without intervention (7,2%)

Parameters that will be measured:

* The effectiveness of Nephrology intervention will be measured giving a punctuation according to the degree of attainment of the objectives. An intervention will be considered effective when a punctuation over 7pt is obtained (adding one point to each of the parameters).
* Routine laboratory tests (baseline and every day after surgery): creatinine, urea, GFR (estimated using the CKD-EPI 10, hemoglobin levels (Hb) and diuresis (mL).
* Parameters at initiation of RRT: serum urea (mmol/L) and serum creatinine (μmol/L), oliguria (defined by urine output <20 mL/h), acidaemia (arterial pH <7.25), K+ (mmol/L), lactic acid
* Duration of RRT (days)
* Number of packed red blood cells, plasma or platelets transfused after the procedure
* Ejection fraction and left ventricular dysfunction 13
* Vascular access used for RRT
* SOFA score

Postoperative day 1 will be defined as the period up to 12pm on the day after surgery, day 2 as the period until 12pm on the subsequent day, and so on.

Statistical analysis An intention-to-treat analysis will be performed considering the results of the patient in the initial assigned group. The outcome data will be measured in all participants (if there is missing data it will be reported and imputed using appropriate methods such as: treating these as if they were observed (e.g. last observation carried forward) Unless otherwise stated, p values and estimates of treatment effects will be based on two-way comparisons.

Continuous variables will be compared between groups using Student's t test or Wilcoxon rank test. Categorical variables will be compared using X2 or Fisher exact test. Subgroup analysis will be performed considering different stages of previous kidney disease and different kind of cardiac surgeries. Survival will be analyzed using Kaplan-Meier and Cox models.

Statistical analysis using SPSS software will be performed.

Ethical issues The trial will be stopped (without one year follow-up) if the in-hospital AKI outcomes are negative (defining that there is more than 25% of differences between groups).

This study has already been approved by the Ethics committee of the Hospital Universitari de Bellvitge on the 10th of July of 2014.

Interim analysis and stopping rules The interim analysis will not be published previously and the stopping rules will be that any patient who do not want to participate in the study, will be dropped-out without any impediment. There will not be an independent data-monitoring committee.

Indemnities: none Publication plan: Results will be published in an international journal. Funder : no funding.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* patients undergoing scheduled cardiac surgery
* Informed consent

Exclusion Criteria:

* a requirement for RRT before surgery
* current outpatient management by a nephrologist or estimated GFR < 45 mL/min/1.73m2 estimated by CKD-EPI equation)
* participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in Acute kidney injury stage defined using KDIGO (Kidney Disease Improving Global Outcomes) criteria | Day of surgery, 4 and 12 months
  rise in serum creatinine ≥26.5 μmol/L in 48 h, or rise 1.5-1.9 times from baseline or Urine output of 0.5 mL/kg/h for 6-12 h

SECONDARY OUTCOMES:
Mortality | through study completion,up to 1 year
  Mortality
Hospitalization days and length of stay in ICU | 1 month
  Hospitalization days and length of stay in ICU
number of participants with Need of Renal Replacement Therapy | 1 month
  Need of Renal Replacement Therapy
number of participants with Anemia and need of blood transfusion | 1, 4 and 12 months
  Anemia and need of blood transfusion
number of participants with Need of Use of inotropes after surgery | The day of surgery
  Use of inotropes after surgery (number, type, dose)
number of participants with Metabolic complications | 4 and 12 months
  Diabetes mellitus, hypertension, dyslipidemia after discharge and hyperuricemia
Estimated glomerular filtration rate | Each day of the hospitalization, 4 and 12 months
  Estimated glomerular filtration rate by CKD-EPI formulae
number of participants with Inflammation adverse events | through study completion, up to 1 year
  Reactive C Protein value

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Montero, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Nephrology Department. Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Codina S, Oliveras L, Ferreiro E, Rovira A, Coloma A, Lloberas N, Melilli E, Hueso M, Sbraga F, Boza E, Vazquez JM, Perez-Fernandez JL, Sabater J, Cruzado JM, Montero N. Nephrology intervention to avoid acute kidney injury in patients awaiting cardiac surgery: randomized clinical trial. Front Nephrol. 2024 Nov 13;4:1470926. doi: 10.3389/fneph.2024.1470926. eCollection 2024. PMID 39606581